CLINICAL TRIAL: NCT04606459
Title: A Multicentric Randomized Open Label Controlled Superiority Trial to Evaluate the Effectiveness of a Therapy With a Coronary Sinus Reducer as Compared to Guideline-directed Medical Therapy in Patients With Refractory Microvascular Angina
Brief Title: COSIMA: COronary SInus Reducer for the Treatment of Refractory Microvascular Angina
Acronym: COSIMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Shockwave Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Tommaso Gori, Clinical Professor, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-15363
Record Dates: First submitted 2020-10-18; First posted 2020-10-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Coronary Microvascular Disease; Refractory Angina
MeSH Terms: conditions — Microvascular Angina; Angina Pectoris

STUDY DESIGN:
Intervention Model Description: In the current randomized, controlled, parallel-groups trial, patients will be randomized to guideline-directed optimal medical therapy with coronary sinus Reducer (Neovasc Reducer™ System) implantation or guideline-directed medical therapy alone.
Masking Description: Given the nature of the intervention, there is not possibility to use a blinded design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimal medical therapy (Active Comparator): Optimal medical therapy consisting of acetyl salicylic acid, statins, beta-blockers, calcium channel-antagonists, ranolazine will be administered at the discretion of the physician as recommended by the most recent European Society of Cardiology (ESC) guidelines.
  Long-acting nitrates will not be administered unless for patients with fractional flow reserve (FFR)<0.8 or with previously reported good response. Short-acting nitrates may be administered in patients in whom concomitant epicardial spasm is suspected, but they have no documented effect on microvascular angina.
  Interventions: Other: Optimal medical therapy
- Coronary sinus reducer (Experimental): The device being studied is the Neovasc Reducer™ System. Each patient in the Reducer group will be implanted with a single Reducer according to the instructions for use.
  Interventions: Device: Coronary sinus reducer

INTERVENTIONS:
Device: Coronary sinus reducer — The Reducer System comprises the Reducer device (Reducer) pre-mounted on the Reducer Balloon Catheter. The Reducer System is available in one model size. The Reducer is a sterile, single-use, implantable device designed to establish a narrowing in the coronary sinus (CS) and is intended to improve perfusion to ischemic myocardium in the presence of reversible ischemic heart disease to alleviate the symptoms of refractory angina. The device is implanted percutaneously through the right internal jugular vein into the CS. The Reducer is pre-mounted (crimped) on the Reducer Balloon Catheter which, after inflation, causes device expansion and apposition with the vessel wall. The balloon catheter is then deflated and removed from the CS, leaving the device permanently implanted.
  Arms: Coronary sinus reducer
Other: Optimal medical therapy — Guideline-directed medical therapy
  Arms: Optimal medical therapy

SUMMARY:
Patients with refractory microvascular angina fulfilling the predefined inclusion and exclusion criteria will be enrolled in this randomized trial. The primary objective is to investigate whether the proportion of patients reporting an improvement in Canadian Cardiovascular Society (CCS) angina class (≥2 classes) is different at six months after implantation of a Coronary Sinus Reducer followed by optimal medical therapy (OMT) compared to OMT alone.

DETAILED DESCRIPTION:
Recent data show that 47% of the patients undergoing coronary angiography for angina have no epicardial disease. Of these, 52% have isolated microvascular angina, 17% have isolated vasospastic angina, 20% have both, and 11% have non-cardiac chest pain. These data suggest that microvascular disease is a highly prevalent condition, which might affect as many as 25% of all patients undergoing coronary angiography (without counting patients with acute coronary syndromes and those with mixed epicardial and microvascular disease). Based on an estimate of the Woman´s Ischemia Syndrome Evaluation (WISE) study, 3-4 million patients with symptoms of myocardial ischemia have non-obstructive coronary artery disease in the United States of America. These patients represent a significant burden in terms of mortality and morbidity as well as in terms of healthcare costs due to disability, hospitalization, and repeat testing.

Patients with microvascular angina require frequent hospitalizations, undergo repeat invasive procedures, have an impaired quality of life and a poor prognosis, since patients with a high index of microvascular resistances) have a higher risk of mortality (hazard ratio (HR) 1.6[0.8-3.4], P<0.001)). An analysis of the WISE study identified an impaired coronary flow reserve in the absence of epicardial disease as the strongest predictor of 5-year adverse events (26.7% versus 12.2%, HR 1.2[1.1.-1.4], P=0.008).

Although its importance is acknowledged by the most recent guidelines, microvascular angina represents a major clinical challenge. In particular, there is a strong disagreement on its classification, on the several mechanisms behind its pathophysiology, and the therapeutic alternatives available remain unsatisfactory.

Despite these uncertainties, there is a consensus that this condition is highly frequent, as it affects up to two-thirds of patients who suffer from stable angina and either have no coronary stenoses at angiography or have combined epicardial and microvascular disease.

The limits of medical therapy Traditional anti-ischaemic drugs are the first step in medical treatment, but their effectiveness is very limited in the setting of microvascular disease. Short-acting nitrates can be used to treat anginal attacks, but since nitrates are only effective on large arteries, this therapy is only indicated for the therapy of patients whose symptoms are caused by spasm of epicardial coronaries, and not for true microvascular angina. Beta-blockers limit myocardial oxygen consumption but do not affect the mechanisms of microvascular disease. Calcium antagonists, have shown variable results in clinical trials, but the limitation of this approach is that a significant heterogeneity exists in the types of calcium channels in the vasculature.

Evidence on the coronary sinus reducer In recent years, the coronary sinus reducer has been introduced to treat refractory angina in patients with refractory angina due to obstructive coronary artery disease (CAD) and no revascularization options, a situation similar to microvascular disease. This novel therapy is based on the concept that an elevation in backward pressure in the coronary venous system provokes dilatation of the subendocardial arterioles, resulting in a significant reduction of vascular resistance in this area and a redistribution of blood flow to these ischaemic subendocardial layers. Numerous studies confirm the efficacy of the Reducer for patients suffering from angina who are not candidates for revascularization. Preliminary evidence supporting the use of this device in microvascular disease patients also exists, but requires confirmation in a large, randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤85 years
* Chronic coronary syndrome (including patients with anginal equivalents) refractory angina CCS class III-IV despite guideline-directed medical therapy
* Evidence of reversible ischemia on non-invasive testing
* Evidence of microvascular disease as diagnosed invasively by at least one of the following:

  1. index of microvascular resistances (IMR) >25 and/or
  2. coronary flow reserve (CFR) <2.0) with fractional flow reserve (FFR)>0.8.
* Willingness to participate and ability to understand, read and sign the informed consent document before enrollment in the trial.

Exclusion Criteria:

Subjects presenting at least one of the following criteria will not be enrolled in the trial

* Recent (within 3 months) acute coronary syndrome
* Recent (within 6 months) revascularization by percutaneous coronary intervention (PCI, stent) or coronary artery by-pass surgery (CABG)
* Recent (within 30 days) unsuccessful PCI
* Decompensated congestive heart failure (CHF) or hospitalization due to CHF during the last 3 months
* Left ventricular ejection fraction of <30%
* Mean right atrial pressure >15mmHg
* Anomalous or abnormal CS anatomy (e.g., tortuosity, aberrant branch, persistent left superior vena cava [SVC]) as demonstrated by angiogram
* CS diameter at the site of planned Reducer implantation greater than 13mm or less than 9.5mm as measured by angiogram
* Severe chronic obstructive pulmonary disease (COPD) indicated by a forced expiratory volume in one second that is less than 55 percent of the predicted value
* Severe valvular heart disease
* A pacemaker electrode in the coronary sinus
* Tricuspid valve replacement or repair
* Chronic renal failure (serum creatinine >2mg/dL), and/or on chronic hemodialysis
* Moribund, or with comorbidities limiting life expectancy to less than one year
* Known severe reaction to required procedural medications
* Known allergy to stainless steel or nickel
* Need for Magnetic Resonance Imaging (MRI) within 8 weeks after reducer implantation
* Contraindication to dual antiplatelet therapy
* Female of childbearing potential (last menstruation within the last 12 months or who did not undergo tubal ligation, ovariectomy or hysterectomy)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2029-10-20 (Estimated)

PRIMARY OUTCOMES:
Change in Canadian Cardiovascular Society angina class by two or more classes | 6 months
  Proportion of patients improving ≥2 CCS angina classes at six months after the implantation followed byoptimal medical therapy (OMT) compared to OMT alone.

SECONDARY OUTCOMES:
Change in angina severity according to the Seattle Angina Questionnaire | Six months
  change in angina severity as assessed by the Seattle Angina Questionnaire (SAQ-7, range from 0 to 100, with 100 as minimal physical limitation and angina and 0 as maximal limitation and angina) at six months.
Number of participants with technical success | Implantation day
  - Technical success: in the Reducer group, defined as successful delivery and deployment of the Reducer to the intended site as assessed by the investigator
Procedural success | Implantation day
  - Procedural success: in the Reducer group, defined as technical success and the absence of acute need for clinically-driven intervention to address an Adverse or Serious Adverse Device Effect prior to hospital discharge, as adjudicated by the Clinical Events Committee (CEC)
Frequency of use of sublingual nitrates (times per week) | 6 months, 1 year, 5 years
  Use of sublingual nitrates
Parameters of angina and quality of life | at 6 months
  Seattle Angina Questionnaire:
  * SAQ-7 Physical limitation scale
  * SAQ-7 angina stability scale
  * SAQ-7 angina frequency scale
  * SAQ-7 quality of life
  * SAQ-7 Treatment Satisfaction
  * Disease perception scale
Incidence of adverse events | 5 years
  Combined incidence of :
  Death (all cause and cardiovascular) Myocardial infarction Revascularization Periprocedural complications
Number of documented Emergency Department (ED) visits due to angina episodes | 6 and 12 months
  Number of documented Emergency Department (ED) visits due to angina episodes
Canadian Cardiovascular Society angina class | 6 months, 1 year, 5 years
  CCS Angina class
Number of unplanned hospitalizations for cardiac ischemia, angina or anginal equivalent, heart failure | 6 months, 1 year, 5 years
  Unplanned hospitalization for cardiac ischemia, angina or anginal equivalent, heart failure
Change in 5-level EQ-5D version (EQ-5D-5L) | 6 months
  5-level EQ-5D version (EQ-5D-5L, EuroQol Group) change in visual score, from 0 to 100 (best)
Beck depression inventory | 6 months
  Beck depression inventory, from 1 (best) to 40 (worst)

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Cardiology, Cardiology I, university hospital Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Upon motivated request all data will be shared